CLINICAL TRIAL: NCT05849584
Title: Levator Hiatal Dimensions and Mode of Delivery
Acronym: LEVDIM
Status: Withdrawn | Type: Observational
Why Stopped: The study will not proceed due to lack of funding.
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 423957
Record Dates: First submitted 2023-01-19; First posted 2023-05-09 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Floor; Rupture; Childbirth Problems; Pelvic Floor Dyssynergia
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

GROUPS / COHORTS (1):
- Pregnant women
  Interventions: Other: Transperineal ultrasound

INTERVENTIONS:
Other: Transperineal ultrasound — A 2D scan will be performed of one experienced clinician. The average of 3 2D levator hiatal anteroposterior measurements will be stored. Then, a 3D/4D ultrasound examination of the pelvic floor will be performed using a Voluson S10, E8 or E10 (GE healthcare, Zipf, Austria) device with a RAB 4-8 MHz curved array transducer with the acquisition angle set at 85 degrees. Offline analysis of the ultrasound volumes will be performed using the 4D view (GE Healthcare, Austria) software, blinded to all clinical data. Hiatal anteroposterior diameter will be measured in both 2D and 3D. Hiatal area and hiatal transverse diameter will be measured in the 3D volume

SUMMARY:
The aim of this observational study is to learn about how muscle dimensions of the pelvic floor measured during pregnancy in primigravida impact birth mecanics and mode of delivery. Tha main aims are to 1. Explore associations between mode of delivery and hiatal dimensions measured by transperineal ultrasound antenatally and 2. Explore the association between duration of 2nd stage of labour and hiatal dimensions.

A pelvic floor ultrasound examination will be performed between pregnancy week 12 and 20 and levator ani muscle hiatal dimensions will be compared between women having a normal vaginal delivery and women with emergency cesarean or operative vaginal deliveries.

DETAILED DESCRIPTION:
The women will be enrolled and examined at the 12-week routine ultrasound examination after informed consent and examined again at the 18 weeks gestation examination. The women will be examined in the supine position on a bed with knees and hips semi-flexed and abducted. Bladder and bowel should be emptied prior to the examination. They will be instructed in how to perform pelvic floor contraction and maximal Valsalva maneuver.

First, a 2D scan will be performed of one experienced clinician. The average of 3 2D levator hiatal anteroposterior measurements will be stored. Then, a 3D/4D ultrasound examination of the pelvic floor will be performed using a Voluson S10, E8 or E10 (GE healthcare, Zipf, Austria) device with a RAB 4-8 MHz curved array transducer with the acquisition angle set at 85 degrees. Offline analysis of the ultrasound volumes will be performed using the 4D view (GE Healthcare, Austria) software, blinded to all clinical data. Hiatal anteroposterior diameter will be measured in both 2D and 3D. Hiatal area and hiatal transverse diameter will be measured in the 3D volume. These measures have previously been demonstrated to have high interrater and intrarater reliability in women in this study population.

Details regarding maternal height, weight, age, ethnicity, marital status, employment, induction of labour, duration of active 2nd stage of labour, gestational length, use of epidural analgesia, indication for operative delivery (slow progress or fetal distress), mode of delivery (forceps, vacuum, cesarean section), infant birthweight, head circumference, Presentation (occiput anterior/ posterior), head station at intervention, infant gender, Apgar score, perineal trauma, postpartum hemorrhage, will be collected from electronic patient journals after delivery. The women will be informed that they may be contacted within 2 years after delivery for a follow up, but separate consent will be needed.

Participants will have a unique study number and the coupling list will be stored on a safe area at St. Olav's server.

ELIGIBILITY:
Inclusion Criteria

* Age over 18 years
* Ability to consent
* Singleton pregnancy

Exclusion criteria

* Previous deliveries > 16 weeks gestation
* Previous pelvic floor surgery
* Anomalies affecting the pelvic floor function (such as myelomeningocele)
* Epilepsy, since this might influence intervention during delivery
* Women with elective cesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 400 nulliparous pregnant women recruited at routine ultrasound scan i nearly pregnancy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | Assessed at 1 day of childbirth
  Normal vaginal, vacuum assisted vaginal, forceps assisted vaginal or emergency cesarean delivery
Levator hiatal dimensions | Measured in pregnancy week 12
  levator hiatal anteroposterior diameter and levator hiatal area at rest measured with 2D and 3D ultrasound
Levator hiatal dimensions | Measured in pregnancy week 18
  levator hiatal anteroposterior diameter and levator hiatal area at rest measured with 2D and 3D ultrasound

SECONDARY OUTCOMES:
Duration of second stage of delivery | Assessed at 1 day of childbirth
  Number of minutes from full dillatation of the cervix until the baby is born
Pernineal tears | Assessed at 1 day of childbirth
  Grade of perineal tear. No tear, grade 1, 2, 3, 4 or deep vaginal tear
Postpartum haemorrage | Assessed at 1 day of childbirth
  Amount in ml of postpartum haemmorage
womans experience of transperineal ultrasound | Assessed at pregnancy week 12 and week 18
  Qualitative assessment of the womans experience of transperineal ultrasound
Interrater validity of ultrasound measurements | Assessed 3 months after childbirth
  For analysis of intrarater reliability for ultrasound measurements, we will use the intraclass correlation coefficient (ICC) two-way mixed effects, absolute agreement model. To determine interrater reliability, we will use the ICC two-way random effects, absolute agreement model, applying both the mean of three raters and single measurements. [20]. The following ICC cut-offs will be applied: < 0.20 = poor reliability, 0.20-0.40 = fair reliability, 0.41-0.60 = moderate reliability, 0.61-0.80 = good reliability and > 0.80 = excellent reliability

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Volløyhaug, PhD, Principal Investigator — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Levanger Sykehus, Levanger
  - st.Olavs hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No